CLINICAL TRIAL: NCT06464991
Title: A Phase III Randomized, Controlled Study of Equecabtagene Autoleucel Injection in Subjects With Lenalidomide-Refractory R/R Multiple Myeloma
Brief Title: A Phase III Study of Eque-cel in Subjects With Len-refractory RRMM (FUMANBA-03)
Acronym: FUMANBA-03
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing IASO Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT103AC004
Record Dates: First submitted 2024-05-30; First posted 2024-06-18 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Eque-cel
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; pomalidomide; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Drug:Equecabtagene Autoleucel Injection
  Interventions: Drug: Equecabtagene Autoleucel Injection
- Control group (Active Comparator): Drug:
  Daratumumab, Bortezomib, Dexamethasone, Pomalidomide, DPd group: Daratumumab, Pomalidomide, Dexamethasone PVd group: Bortezomib, Dexamethasone, Pomalidomide
  Interventions: Drug: Daratumumab; Drug: Pomalidomide; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Equecabtagene Autoleucel Injection — dosage form: injection, dosage: 1.0×10^6 CAR-T/kg, frequency: single dose.
  Other Names: FUCASO
  Arms: Experimental group
Drug: Daratumumab — dosage form: Injection dose level:16mg/kg frequency: 28days/cycle for DPd regimen
  * Cycle1-2：D1, D8, D15, D22；
  * Cycle3-6：D1, D15；
  * above Cycle7：D1
  Arms: Control group
Drug: Pomalidomide — dosage form:capsule. doseage form: capsule. dose level: 4mg/d. frequency: every cycle: D1-D21 for DPd regimen, D1-D14 for PVd regimen.
  Arms: Control group
Drug: Bortezomib — dosage form: subcutaneous injection. dose level: 1.3mg/m2. frequency: 21days/cycle for PVd regimen cycle 1-8: D1,D4, D8, D11； above cycle 9: D1, D8.
  Arms: Control group
Drug: Dexamethasone — dosage form: oral or intravenus injection. dose level:20mg/d. frequency: for DPd: every cycle, D1, D2, D8, D9, D15, D16, D22, D23； for PVd: Cycle1-8：D1, D2, D4, D5, D8, D9, D11, D12; above Cycle 9: D1, D2, D8, D9.
  Arms: Control group

SUMMARY:
This is a multicenter, randomized, controlled, open-label, phase III clinical study to evaluate the efficacy of Equecabtagene Autoleucel Injection versus standard therapy in subjects with lenalidomid-refractory RRMM who have received 1-2 lines of prior therapy.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a malignant neoplasm of plasma cells that accounts for more than 10%-20% of hematologic malignancies worldwide, leading to marrow failure and bone destruction. Equecabtagene Autoleucel (eque-cel) is an autologous chimeric antigen receptor T-cell (CAR-T) therapy that targets B-cell maturation antigen (BCMA), which expressed on both mature B lymphocytes and malignant plasma cells. The primary objective for this study is to compare the efficacy of eque-cel versus standard therapy in lenalidomid-refractory RRMM. Subjects will undergo screening with informed consent. After enrollment, randomization will be conducted followed by study treatment in experimental or control group. A follow-up phase will include assessments for safety, efficacy evaluation and pharmacokinetics monitoring (experimental arm) . The duration of this trial is about 6 years.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years of age (inclusive of critical values), either gender.
2. The subject was previously diagnosed with multiple myeloma and had received 1-2 lines of therapy (including chemotherapy regimens based on proteasome inhibitors and immunomodulatory agents, with each line of therapy receiving at least 1 full cycle ; Documented disease progression during or within 12 months after the most recent anti-myeloma therapy.
3. Subjects was lenalidomide-refractory during prior therapy.
4. ECOG score of 0 or 1.
5. Subjects must have appropriate organ function and meet all of the following laboratory test results before enrollment:

(1) Haematology: absolute neutrophil count (ANC) ≥1×10^9/L (support with growth factor is allowed, but must not have received supportive treatment within 7 days before the laboratory test); Absolute lymphocyte count (ALC) ≥0.3×10^9/L; Platelets ≥50×10^9 / L (must not have received platelet transfusion within 7 days prior to laboratory test); Hemoglobin ≥60g/L (must not have received red blood cells transfusion within 7 days prior to laboratory test); (2) Hepatic function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times of upper limit of normal (ULN); Serum total bilirubin ≤1.5 times of ULN; (3) Renal function: creatinine clearance (CrCl) calculated by Cockcroft-Gault formula ≥ 40 ml/min; (4) Coagulation: fibrinogen≥1.0 g/L; activated partial thromboplastin time (APTT) ≤ 1.5×ULN, pro-thrombin time (PT) ≤ 1.5 × ULN; (5) Pulse oxygen saturation > 91%; (6) Left ventricular ejection fraction (LVEF)≥50%;

6. Subjects agree to use effective tools or drug contraception (excluding safe period contraception) after signing the informed consent form.

7. Subjects must agree to sign or personally sign an ethics committee-approved informed consent form before starting any screening procedures.

Exclusion Criteria:

1. Subjects who have used or required long-term immune-suppressive agents (e.g., cyclosporine or systemic steroids) within 14 days prior to enrollment, but the use of physiological substitutes, intermittent, topical, and inhaled steroids is allowed.
2. Subjects who have undergone autologous haematopoietic stem cell transplantation (Auto-HSCT) within 12 weeks prior to randomization, or who have previously undergone allogeneic haematopoietic stem cell transplantation (Allo-HSCT).
3. Subjects received the following anti-tumor treatments before enrollment: (1)Treated with an immunomodulator within 7 days, or; (2)Received plasma exchange, radiotherapy (except local radiotherapy for myeloma-related bone lesions), cytotoxic chemotherapy, treatment with proteasome inhibitors or other investigational drug within 14 days, or; (3) Treatment with monoclonal antibody for multiple myeloma within 21 days, or; (4) Received other anti-cancer therapy within 14 days or at least 5 half-lives (whichever is shorter) prior to enrollment.
4. Significant cardiac disorder.
5. Unstable systemic disease as judged by the investigator: including but not limited to severe liver, renal, or metabolic disease requiring medication.
6. The subject will not be able to participate in this study if the investigator determines that the subject meets any of the following conditions: (1) Subjects with a history of allergic reaction to the excipient components (DMSO and albumin) of Eque-cel, fludarabine, cyclophosphamide, tocilizumab, or; (2) Subjects who are intolerant to dexamethasone, or; (3) Subjects who have a Life-threatening allergy, hypersensitivity reaction, or intolerance to pomalidomide and/or its excipients (intolerance is defined as discontinuation of prior treatment due to any AE related to pomalidomide) or;
7. Have malignancies other than multiple myeloma within 5 years before screening, excluding cervical carcinoma in situ after radical surgery, basal cell or squamous cell skin cancer, localized cancer of prostate after radical prostatectomy, breast ductal carcinoma in situ after radical mastectomy or carcinoma papillary thyroid after radical thyroidectomy.
8. Subjects suspected or confirmed to have central nervous system involvement of MM during the screening period.
9. Subjects with concurrent plasma cell leukemia(defined as plasma cell proportion in peripheral blood > 5%), Waldenström macroglobulinaemia, POEMS syndrome (polyneuropathy, organ hypertrophy, endocrinopathy, monoclonal protein and skin changes) or primary amyloidosis during screening period.
10. Have extramedullary multiple myeloma-extraosseous (EM-E); have multiple extramedullary multiple myeloma-bone related (EM-B) and the maximum transverse diameter of any lesion is >3cm; have a single EM-B and the maximum transverse diameter of the lesion is >3cm.
11. Had major surgery within 2 weeks prior to randomization or planned to have surgery within 2 weeks after study treatment (except for subjects who were scheduled to have surgery under local anesthesia).
12. Subject with uncontrollable infection.
13. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and hepatitis B virus (HBV) DNA quantification in peripheral blood was higher than the lower limit of detection; hepatitis C virus (HCV) antibody positive and hepatitis C virus (HCV) RNA positive in peripheral blood; Human immunodeficiency virus (HIV) antibody positive; Syphilis test positive; positive cytomegalovirus (CMV) DNA.
14. Pregnant or breastfeeding women.
15. The subject has a history of central nervous system disorder within 6 months prior to signing the informed consent form.
16. Non-hematological toxicity reactions due to prior treatment have not resolved to baseline or ≤ Grade 1 (NCI-CTCAE v5.0, alopecia, Grade 2 peripheral neuropathy were excepted).
17. Subjects had other conditions that the investigator considered unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) as assessed by Independent Review Committee (IRC) | up to 5 years from randomization
  The time from randomization to the first documented disease progression as determined by IRC or death due to any cause

SECONDARY OUTCOMES:
Minimal Residual Disease (MRD) negativity rate at 12 months | up to 5 years from randomization
  The proportion of subjects who achieve MRD negativity (using next-generation flow cytometry according to EuroFlow standard operating procedures) and complete response (CR) or better, as assessed by IRC, 12 months (±3 months) post-randomization
Overall MRD negativity rate | up to 5 years from randomization
  The proportion of subjects who achieve MRD negativity at any time after the date of randomization and before the initiation of subsequent therapy
Duration of MRD negativity | up to 5 years from randomization
  The time from first achievement of MRD negativity to the first subsequent positive MRD status
Complete Response Rate（CRR） | up to 5 years from randomization
  The proportion of subjects who achieve CR or better post-randomization among all randomized subjects
Very good partial response or better response (≥VGPR) rate | up to 5 years from randomization
  The proportion of subjects who achieve sCR, CR, or VGPR post-randomization among all randomized subjects
Overall Response Rate（ORR） | up to 5 years from randomization
  The proportion of subjects who achieve sCR, CR, VGPR, or PR post-randomization among all randomized subjects.
Duration of Response (DOR) | up to 5 years from randomization
  The time from the first date of initial documented response (≥PR) to the date of first disease progression or death from any cause, whichever occurs first, post-randomization
Event-Free Survival (EFS) | up to 5 years from randomization
  Time from randomization to the first occurrence of any of the following events: death, disease progression, initiation of a new anti-myeloma therapy, addition of other treatments, or occurrence of fatal or intolerable adverse effects
Overall Survival（OS） | up to 5 years from randomization
  Defined as the time from randomization to death due to any cause
Time to Next Treatment（TTNT） | up to 5 years from randomization
  Time from randomization to the initiation of a new subsequent anti-myeloma therapies
Incidence of Adverse events | up to 5 years from randomization
  Safety Endpoint
Pharmacokinetic Endpoint-Cmax | up to 5 years from Eque-cel infusion
  The maximum concentration (Cmax) of CAR VCN and BCMA CAR-T in peripheral blood after CAR-T infusion
Pharmacokinetic Endpoint-Tmax | up to 5 years from Eque-cel infusion
  the time for CAR VCN and BCMA CAR-T to reach the maximum concentration (Tmax) after CAR-T infusion
Pharmacokinetic Endpoint-AUC | up to 5 years from Eque-cel infusion
  Area under the curve of 29, 85, 169 days and the last time point of PK detection (AUC0-29d, AUC0-85d, AUC0-169d, AUC0-last) for CAR VCN; Area under the curve of 29 days (AUC0-29) for BCMA CAR-T.
Pharmacodynamic Endpoint | up to 5 years from Eque-cel infusion
  The concentration of soluble BCMA in peripheral blood of experimental group at each time point
Health Related Quality of Life Endpoint | up to 5 years from randomization
  Symptoms, function, and overall HRQoL were collected using the validated Patient-Reported Outcomes (PRO) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gui Lu Qiu, PhD, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences; Zhen Cai, PhD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (28):
- China (28):
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing
  - Beijing GoBoard Boren Hospital, Beijing
  - Fu Xing Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - People's Hospital of Peking University, Beijing
  - The first hospital of Jilin University, Changchun
  - West China School of Medicine, West China Hospital of Sichuan University, Chengdu
  - Xinqiao Hospital of AMU, Chongqing
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Sun Yat-sen University Cancer Centre, Guangzhou
  - Zhujiang Hospital of Southern Medical University Guangdong, Guangzhou
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou
  - The Second Affiliated Hospital,Zhejiang University School of Medicine, Hangzhou
  - Qilu Hospital of Shangdong University, Jinan
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Affiliated Drum Tower Hospital, Medical School of Nanjing University, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - The Affiliated People's Hospital of Ningbo University, Ningbo
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjing
  - Tianjin Medical University General Hospital, Tianjing
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Henan Cancer Hospital Affilated Cancer Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No